CLINICAL TRIAL: NCT04321421
Title: Plasma From Donors Recovered From New Coronavirus 2019 As Therapy For Critical Patients With Covid-19
Brief Title: Hyperimmune Plasma for Critical Patients With COVID-19
Acronym: COV19-PLASMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: OSPEDALE CARLO POMA ASST MANTOVA (Unknown)
Responsible Party: Principal Investigator, Cesare Perotti, Head, Immunohematology & Transfusion Service, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRCCSSanMatteoH
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
Keywords: hyperimmune plasma; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Intervention Model Description: Longitudinal assessment of COVID-19 patients treated with hyperimmune plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treated (Experimental): treated with hyperimmune plasma
  Interventions: Other: hyperimmune plasma

INTERVENTIONS:
Other: hyperimmune plasma — administration of hyperimmune plasma at day 1 and based on clinical response on day 3 and 5

SUMMARY:
The outbreak of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), has become pandemic. To date, no specific treatment has been proven to be effective. Promising results were obtained in China using Hyperimmune plasma from patients recovered from the disease.The investigators plan to treat critical Covid-19 patients with hyperimmune plasma.

DETAILED DESCRIPTION:
Apheresis from recovered donors will be performed with a cell separator device , with 500-600 mL of plasma obtained from each donor. Donors are males, age 18 yrs or more, evaluated for transmissible diseases according to the italian law. Adjunctive tests will be for hepatitis A virus, hepatitis E virus and Parvovirus B-19. All donors will be tested for the Covid-19 neutralizing title. Each plasma bag obtained from plasmapheresis will be immediately divided in two units and frozen according to the national standards and stored separately.

Based on experience published in literature 250-300 mL of convalescent plasma will be used to treat each of the recruited patients at most 3 times over 5 days.

ELIGIBILITY:
Inclusion Criteria:

* age >=18 yrs
* positive for reverse transcription polymerase chain reaction (RT-PCR) severe acute respiratory syndrome (SARS)-CoV-2
* Acute respiratory distress syndrome (ARDS) moderate to severe, according to Berlin definition, lasting less than10 days
* Polymerase chain reaction (PCR) increased by 3.5 with respect to baseline or >1.8 mg/dl
* need for mechanical ventilation or continuous positive airway pressure (CPAP)
* signed informed consent unless unfeasible for the critical condition

Exclusion Criteria:

* Moderate to severe ARDS lasting more than 10 days
* proven hypersensitivity or allergic reaction to hemoderivatives or immunoglobulins
* consent denied

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
death | within 7 days
  death from any cause

SECONDARY OUTCOMES:
time to extubation | within 7 days
  days since intubation
length of intensive care unit stay | within 7 days
  days from entry to exit from ICU
time to CPAP weaning | within 7 days
  days since CPAP initiation
viral load | at days 1, 3 and 7
  naso-pharyngeal swab, sputum and BAL
immune response | at days 1, 3 and 7
  neutralizing title

CONTACTS AND LOCATIONS:
Overall Officials: Cesare Perotti, MD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo di Pavia
Locations (2):
- Italy (2):
  - Catherine Klersy, Pavia, PV
  - Ospedale Asst Carlo Poma Mantova, Mantova

IPD SHARING:
Plan to Share IPD: Undecided
will be decided

REFERENCES:
- [Background] Chen L, Xiong J, Bao L, Shi Y. Convalescent plasma as a potential therapy for COVID-19. Lancet Infect Dis. 2020 Apr;20(4):398-400. doi: 10.1016/S1473-3099(20)30141-9. Epub 2020 Feb 27. No abstract available. PMID 32113510
- [Background] WHO. Clinical management of severe acute respiratory infection when novel coronavirus (nCoV) infection is suspected. 2020. https://www.who. int/docs/default-source/coronaviruse/clinical-management-of-novel-cov. pdf (accessed Feb 20, 2020).
- [Background] Lai ST. Treatment of severe acute respiratory syndrome. Eur J Clin Microbiol Infect Dis. 2005 Sep;24(9):583-91. doi: 10.1007/s10096-005-0004-z. PMID 16172857
- [Background] WHO. Use of convalescent whole blood or plasma collected from patients recovered from Ebola virus disease for transfusion, as an empirical treatment during outbreaks. 2014. http://apps.who.int/iris/rest/ bitstreams/604045/retrieve (accessed Feb 20, 2020).
- [Background] Arabi Y, Balkhy H, Hajeer AH, Bouchama A, Hayden FG, Al-Omari A, Al-Hameed FM, Taha Y, Shindo N, Whitehead J, Merson L, AlJohani S, Al-Khairy K, Carson G, Luke TC, Hensley L, Al-Dawood A, Al-Qahtani S, Modjarrad K, Sadat M, Rohde G, Leport C, Fowler R. Feasibility, safety, clinical, and laboratory effects of convalescent plasma therapy for patients with Middle East respiratory syndrome coronavirus infection: a study protocol. Springerplus. 2015 Nov 19;4:709. doi: 10.1186/s40064-015-1490-9. eCollection 2015. PMID 26618098
- [Background] Hung IF, To KK, Lee CK, Lee KL, Chan K, Yan WW, Liu R, Watt CL, Chan WM, Lai KY, Koo CK, Buckley T, Chow FL, Wong KK, Chan HS, Ching CK, Tang BS, Lau CC, Li IW, Liu SH, Chan KH, Lin CK, Yuen KY. Convalescent plasma treatment reduced mortality in patients with severe pandemic influenza A (H1N1) 2009 virus infection. Clin Infect Dis. 2011 Feb 15;52(4):447-56. doi: 10.1093/cid/ciq106. Epub 2011 Jan 19. PMID 21248066
- [Background] Holshue ML, DeBolt C, Lindquist S, Lofy KH, Wiesman J, Bruce H, Spitters C, Ericson K, Wilkerson S, Tural A, Diaz G, Cohn A, Fox L, Patel A, Gerber SI, Kim L, Tong S, Lu X, Lindstrom S, Pallansch MA, Weldon WC, Biggs HM, Uyeki TM, Pillai SK; Washington State 2019-nCoV Case Investigation Team. First Case of 2019 Novel Coronavirus in the United States. N Engl J Med. 2020 Mar 5;382(10):929-936. doi: 10.1056/NEJMoa2001191. Epub 2020 Jan 31. PMID 32004427
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub6. PMID 37162745
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 Feb 1;2(2):CD013600. doi: 10.1002/14651858.CD013600.pub5. PMID 36734509
- [Derived] Piechotta V, Iannizzi C, Chai KL, Valk SJ, Kimber C, Dorando E, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2021 May 20;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub4. PMID 34013969
- [Derived] Chai KL, Valk SJ, Piechotta V, Kimber C, Monsef I, Doree C, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2020 Oct 12;10:CD013600. doi: 10.1002/14651858.CD013600.pub3. PMID 33044747
- [Derived] Piechotta V, Chai KL, Valk SJ, Doree C, Monsef I, Wood EM, Lamikanra A, Kimber C, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2020 Jul 10;7(7):CD013600. doi: 10.1002/14651858.CD013600.pub2. PMID 32648959
- [Derived] Perotti C, Del Fante C, Baldanti F, Franchini M, Percivalle E, Vecchio Nepita E, Seminari E, De Silvestri A, Bruno R, Klersy C. Plasma from donors recovered from the new Coronavirus 2019 as therapy for critical patients with COVID-19 (COVID-19 plasma study): a multicentre study protocol. Intern Emerg Med. 2020 Aug;15(5):819-824. doi: 10.1007/s11739-020-02384-2. Epub 2020 May 28. PMID 32468508